CLINICAL TRIAL: NCT03608761
Title: Comparison Between Rebamipide 2% Versus Autologous Serum in the Treatement of the Moderate to Severe Dry Eye Associate With Sjögren Syndrome. Pilot, Crossed, Controled, Randomized And Open Study
Brief Title: Comparison Between Rebamipide 2% Versus Autologous Serum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 055LuPeSo/15
Record Dates: First submitted 2018-07-09; First posted 2018-08-01 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Dry Eye Syndromes; Sjögren Syndrome
Keywords: dry eye; Sjögren syndrome; Rebamipida 2%; autologous serum
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome | interventions — rebamipide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rebamipide 2% (Experimental): 1. - wash-out: 2 weeks
  2. - rebamipide 2% four times a day for 3 months
  3. - controls will be taken at day zero, 30 and 90.
  4. - wash-out: 2 weeks
  5. - autologous serum for 3 months
  Interventions: Drug: Rebamipide
- Autologous serum (Experimental): 1. - wash-out: 2 weeks
  2. - autologous serum four times a day for 3 months
  3. - controls will be taken at day zero, 30 and 90.
  4. - wash-out: 2 weeks
  5. - rebamipe 2% for 3 months
  Interventions: Biological: autologous serum
- autologous serum and rebamipide 2% (Experimental): rebamipide 2% and autologous serum four times a day for 3 months separately by 1 minute between each other controls will be taken at day zero, 30 and 90. this group will not be crossed
  Interventions: Other: autologous serum and rebamipide 2%

INTERVENTIONS:
Drug: Rebamipide — rebamipide 2%
  Other Names: GR
  Arms: Rebamipide 2%
Biological: autologous serum — AS for 3 months
  Other Names: GSA
  Arms: Autologous serum
Other: autologous serum and rebamipide 2% — rebamipide and autologous serum for 3 months
  Other Names: GSAR
  Arms: autologous serum and rebamipide 2%

SUMMARY:
Two-period, controlled, randomized and open clinical trial. The sample was composed of adult women with moderate to severe hypo secretory dry eye associated with Sjögren's syndrome, who attended the ocular surface office, derived from the general ophthalmology clinic, from the Rheumatology or Immunology department. The three interventions were randomized: autologous serum (GSA), Rebamipida 2% (GR) and a combined treatment (GSAR). The following were used as outcome measures: OSDI self-administered questionnaire (Ocular Surface Disease Index), tear-rupture time (BUT), fluorescein staining, Bengal Rose staining and Schirmer's test without anesthesia to assess the answer to each treatment

DETAILED DESCRIPTION:
After having borrowed to participate in the study, we proceeded to the random assignment of each intervention as follow: the last 2 numbers of the clinical history, typical of the ocular surface office, were taken and they were placed in a list in order of lower to higher. Then, each of them was assigned to a number from a table of random numbers. The list was rearranged from lowest to highest using the assigned random number. Finally, the treatment was assigned by simple randomization without replacement. In this way, the subject with the lowest random number, the correspondence in the first treatment drawn. It was continued in the same way, respecting the order assigned by random numbers until completing the 21 subjects.

Three groups of 7 subjects each were formed in this way: treatment group or group Rebamipida (GR); standard treatment group or autologous serum group (GSA) and mixed group or serum and Rebamipide group (GSAR).

Before beginning with the assigned treatment, all the participants was started a period of wash-out of any medicine they were ussing, that least for two weeks. The participants were asked to suspend all the drops that they been used until then (antibiotics, corticosteroids, cyclosporine, artificial tears, autologous serum, etc.), and to place them using only artificial tears (sodium carboxymethyl cellulose). 1%, AUCIC 1%) four times a day in all cases. The purpose was to minimize the effect of the medication that could interfere with the results obtained from the treatments tested. The two week period also allowed the hemotherapy service to prepare the autologous serum for the subjects assigned to this group and initiate the treatment without delays.

Immediately after the washout period, the subjects began to receive the last treatments for 90 days.

After the first intervention cycle and with the objective of influencing the treatment cycle of the first treatment cycle, a second washing period of two weeks duration was carried out.

With the intention of increasing the sample size, the GR and GSA groups were crossed, in this way the patients received the opposite treatment to the start. The second treatment period lasted 90 days, equal to the first.

The mixed group (GSAR) did not cross, ending their participation at the end of the 90 days.

Admission and control of all patients on days 0, 30 and 90 of both cycles were performed by the same ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Sjögren's syndrome
* dry eye symtoms

Exclusion Criteria:

* history of ocular surface surgery less than one year or intraocular surgery less than three months in one or both eyes
* chronic use of drops in one of both eyes (e.g. : treatment for glaucoma)
* anterior segment disease (ocular scar pemphigoid, Stenvens Jhonson syndrome)
* presence of punctung plug (lacrimal plug) inserted in one or both lower lacrimal points
* systemic viral infections (Hepatitis B, Hepatitis C, HIV)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
OSDI | through study completion, an average of 7 months
  ocular surface disease index

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Fa Ross, MD, Principal Investigator — Hospital Nacional Profesor Alejandro Posadas
Locations (1):
- Hospital Nacional Profesor A. Posadas, El Palomar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No